CLINICAL TRIAL: NCT05487365
Title: Implementation and Cost-evaluation of a Smartphone-based Telemonitoring and Digital Support Platform in Patients With Heart Failure: the Bedicare-HF Multicentre Trial
Brief Title: Implementation and Cost-evaluation of a Smartphone-based Telemonitoring and Digital Support in Patients With HF
Acronym: BEDICARE-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Comunicare Solutions SA (Industry)
Collaborators: Jessa Hospital (Other); Hasselt University, Faculty of Medicine and Life Sciences, Hasselt, Belgium (Unknown); KU Leuven (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BEDICARE-HF
Record Dates: First submitted 2022-07-12; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: heart failure; digital support; smartphone; digital health; implementation; remote patient management; telemonitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Eligible patients are consecutive patients that are hospitalised for HF decompensation. All eligible patients will be offered to participate. At the time of inclusion, patients must be in NYHA class II to IV with a LVEF of ≤50%. A total of 330 patients will be included over 6 month. 11 hospitals in Belgium with an HF clinic employing at least one certified HF nurse will be participating in patient recruitment. Patients are not randomised and will all be participating in the smartphone digital support intervention.
  165 patients will be included to use Comunicare app. Patients refusing use Comunicare app will be asked to complete a quality of life (QOL)-questionnaire at 0, 6, and 12 months. A total of 165 patients (who do not want to use the app) will be asked to answer this questionnaire.
  So the app will be made available to 165 patients for home monitoring and another group of 165 patients without an application will be asked to answer quality of life questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with application (Experimental): Eligible patients are consecutive patients that are hospitalised for HF decompensation. The patients will be included in the programme during their hospitalisation or up to one month after hospitalisation. All eligible patients will be offered to participate. At the time of inclusion, patients must be in NYHA class II, III, or IV with a left ventricular ejection fraction (LVEF) of ≤50%. A total of 165 patients with app will be included over 6 month. Patients are not randomised and will all be participating in the smartphone digital support intervention.
  Patients are not randomised and will all be participating in the smartphone digital support intervention.
  So the app will be made available to 165 patients for home monitoring and another group of 165 patients without an application will be asked to answer quality of life questionnaires.
  Patients who agree to use the application can continue to use it after the study, if they wish.
  Interventions: Device: Comunicare Solutions Smartphone Application
- Patients without application (Active Comparator): Patients refusing participation will also be asked to complete a quality of life (QOL)-questionnaire at 6 months and 12 months which will be answered online. A total of 165 patients (who do not want to participate) will be asked to answer this questionnaire.
  So the app will be made available to 165 patients for home monitoring and another group of 165 patients without an application will be asked to answer quality of life questionnaires.
  Patients who agree to use the application can continue to use it after the study, if they wish.
  Interventions: Other: Completing a quality of life (QOL)-questionnaire

INTERVENTIONS:
Device: Comunicare Solutions Smartphone Application — The Comunicare patient support solution is specifically designed for digital support of HF. It consists of an application for patients and a dashboard for the caregivers. The application is a class 1 certified medical device. It includes different modules for patient education, medication adherence, symptoms tracking, electronic patient-reported outcome (ePRO), appointments, and video consultation. Caregiver dashboard application: this web-based application enables caregivers to administrate the care flow and review all patient-reported data and the alarm generated by the system. Security and Privacy: the application complies with strict security and privacy-related regulations. All data storages are encrypted on the patients' smartphone and a server located in an ISO-certified data center located in Belgium, and all information exchanges are highly secured. A GDPR-compliant privacy notice defines how patient personal data is processed and how data protection principles are applied.
  Arms: Patients with application
Other: Completing a quality of life (QOL)-questionnaire — Patients refusing to use Comunicare app will also be asked to complete a quality of life (QOL)-questionnaire at 0, 6 and 12 months which will be answered online.
  Arms: Patients without application

SUMMARY:
The BEDICARE-HF study aims to go further in the research on digital support. The objectives of this study are to demonstrate the feasibility, acceptability, adoption, sustainability and safety of a of a smartphone-based digital support system in the Belgian healthcare system. It also aims to effectiveness, evaluate the cost of implementation of the system and demonstrate the cost-effectiveness.

The study is multi-center, involving the principal investigator, Dr. Pouleur at Cliniques University Clinics Brussels, and co-investigators from 10 hospitals across Belgium. These physicians will enroll 15 patients on Comunicare's online platform. The patients will then have access to the Comunicare application for 6 months, where they will be asked to answer questionnaires and take their vital parameters. They will also have access to documentation on their pathology and will be able to perform videoconferences with their doctor/nurse via the platform.

Eligible patients are patients discharged from hospital for cardiac decompensation. At the time of inclusion, patients must be in NYHA (New-York Heart association) class II, III, or IV, with an LVEF (ejection fraction ejection fraction) of ≤50%.

The BEDICARE-HF project is based on the standard of care that an HF (heart fealure) patient would receive without being part of any study. No other invasive interventions are additionally planned by the project. The patient data collected by the recruiting physician is secured by Comunicare. These fully anonymized data will be sent to Jessa at the end of the study for statistical and economic economic analysis of the results.

The BEDICARE-HF study will therefore investigate the implementation of a digital support intervention for HF supported by smartphone in a European legislative framework. This study will allow further in the evaluation of digital support for HF and to evaluate a low-cost smartphone solution. The results of this study will demonstrate whether and how a smartphone-based digital support system improves self-care capabilities, clinical management, and health outcomes of patients with HF. They will provide important information on the implementation of a implementation of a digital support system in a specific healthcare setting.

DETAILED DESCRIPTION:
Heart failure (HF) is a chronic condition and one of the most challenging issues is to reduce hospital admission and readmission rates for worsening HF. The prevalence of HF is estimated at 1-2% of the total population and ≥10% among people >70 years of age. Increasingly, telemonitoring is used as a solution to intervene at the start of an HF decompensation before the patient starts to be symptomatic and to avoid hospitalization. In recent years, many trials have been published that investigate the utility of telemonitoring in HF in different modalities including invasive monitoring and non-invasive monitoring.

The most recent large randomized controlled trial (RCT) that demonstrated the efficacy of telemonitoring in HF is the TIM-HF2 trial in which a structured remote patient management intervention reduced the percentage of days lost to unplanned cardiovascular hospital admission and all-cause mortality in patients with New York Heart Association (NYHA) class II-III HF with a hospitalization within the last 12 months.

The utility of smartphone applications for patient care is increasingly being appreciated and in Europe, clear guidelines exist for developers who aim to develop software as a medical device. The advantage of using smartphone applications is that little specialized equipment is needed and, if a digital support program is proven successful, implementation can be widely performed at low cost.

In the context of the Covid-19 pandemic, HF patients are particularly suffering from the difficulty to meet their cardiologist and HF nurse on a regular basis. Developing the possibility for remote monitoring is a key alternative to avoid re-hospitalization or severe clinical cardiovascular outcome.

The sponsor present the design of the Bedicare-HF trial, which aims to take digital support research a step further. It uses an implementation design approach in which a real-life setting will be approximated. The trial aims thus to not only demonstrate the effectiveness of a smartphone-based HF digital support approach but also the feasibility of implementation in a European healthcare context. Also, it aims to evaluate the cost-effectiveness of a smartphone-based digital support approach.

Objectives:

The objectives of this study are to demonstrate feasibility, acceptability, adoption, sustainability, and safety of a smartphone-based digital support system in the healthcare system in Belgium and to demonstrate effectiveness, to evaluate the implementation cost of the system, and to demonstrate cost-effectiveness.

Methods:

Study design:

The study design is a multicenter implementation trial. The conduct of the study is guided by good clinical practice (GCP) in accordance with the Declaration of Helsinki and the laws and regulations applicable in Belgium. Written approval from the Ethics Committees at all involved centers is required and informed consent must be provided by each patient.

Patient recruitment:

Eligible patients are consecutive patients that are hospitalized for HF decompensation. The patients will be included in the program during their hospitalization or up to one month after hospitalization. All eligible patients will be offered to participate. At the time of inclusion, patients must be in New York Heart Association (NYHA) class II, III, or IV with a left ventricular ejection fraction (LVEF) of ≤50%. A total of 330 patients will be included over 6 month. In total, 11 hospitals (local investigators) in Belgium with an HF clinic employing at least one certified HF nurse will be participating in patient recruitment. Patients are not randomized and will all be participating in the smartphone digital support intervention.

A screening register will be kept including reasons why eligible patients that do not participate are disregarding inclusion. Patients refusing app using will also be asked to complete a quality of life (QOL)-questionnaire at 6 months and 12 months which will be answered online. A total of 165 patients (who do not want to use the app) will be asked to answer this questionnaire.

So the app will be made available to 165 patients for home monitoring and another group of 165 patients without an application will be asked to answer quality of life questionnaires.

Patients who agree to use the application can continue to use it after the study, if they wish.

Digital support platform The digital support intervention uses the Comunicare patient support solution specifically designed for digital support of HF. The solution consists of a smartphone-based mobile application designed to be used by patients and a web-based dashboard application to be used by the caregivers. The application is a class 1 certified medical device. It includes different modules for patient education, medication adherence, tracking of vital signs and symptoms, electronic patient-reported outcome (ePRO), appointments, and video consultation.

Patient Education module: a knowledge base has been configured into the application to provide patients with information about HF based on the latest ESC guidelines and the local reimbursement context. The patient information that is provided includes descriptions of the function of the heart, the causes of HF, and advice about how to self-manage and understand HF.

Medication adherence: the application enables patients to maintain a medication list and to configure a reminder system to receive notifications. If medication is not taken an explanation for non-intake can be provided.

Tracking of vital signs and symptoms: the application enables patients to track and input vital signs and symptoms as recommended by the caregivers. A notification can be configured to remind the moment of measurement. Measured values can be inserted manually or captured directly from validated connected devices (blood pressure monitor, weight scale, activity tracker). Alarm limits can be set, and an alarm will then be triggered as soon as an input breaches the alarm limit. A Bluetooth-compatible blood pressure monitor and weighing scale will be provided at inclusion. If preferred by the patient manual input through their own devices can be performed.

Electronic patient-reported outcome (ePRO): the application enables patients to complete questionnaires about their QOL. A notification can be configured to remind the moment to fill the questionnaires. When available, scoring of the questionnaires is generated in the dashboard for caregivers.

Appointments and video consultation: the application includes an electronic agenda that can be input manually by the patients or automatically synchronized with the hospital system. It also includes a secure video consultation that can be triggered by the caregivers when deemed necessary after reviewing the patient-reported data.

Caregiver dashboard application: this web-based application enables caregivers to administrate the care flow and review all patient-reported data and the alarm generated by the system.

Security and Privacy: the application complies with strict security and privacy-related regulations. All data storages are encrypted on the patients' smartphone and a server located in an ISO-certified data centre located in Belgium, and all information exchanges are highly secured. A General Data Protection Regulation (GDPR)-compliant privacy notice defines how patient personal data is processed and how data protection principles are applied.

According to the General Personal Data Regulation (GPDR), the data controller determines the purposes for which and the means by which personal data is processed and the data processor processes personal data only on behalf of the controller. The duties of the processor towards the controller are specified in a contract agreement and a Data Processing Agreement (DPA).

In the context of a normal usage of the application, the hospital is data controller and Comunicare Solutions SA is the data processor.

However, in the context of the clinical study, Comunicare Solutions SA is subject to the rights and obligations as "data controller" set forth under the GDPR in relation to the processing of personal data for the purpose of conducting the Study in accordance with the Protocol. In that respect Comunicare Solutions SA shall be considered as data controller of all Personal Data processed specifically for Study purposes.

Each participating center is subject to the rights and obligations as "data processor" set forth under the GDPR in relation to the processing of personal data for the purpose of conducting the Study in accordance with the Protocol.

Each participating center is also subject to the rights and obligations as a separate "data controller" set forth under the GDPR in relation to the processing of personal data of its patients for purposes other than conducting the Study. In particular, each participating center remains data controller of the data contained in the patients' medical records for the purposes of providing medical care to its patients and for academic research purposes.

Comunicare Solutions SA will provide patients with a GDPR policy, as required to inform the patient about his/her rights related to their personal data. The hospital will provide the patients with an informed consent document.

Comunicare Solutions SA will provide each participating center an appropriate number of patient access cards. Each patient access card displays an anonymous user ID and password as well as a scannable QR code (quick response code) . Once the written informed consent form (ICF) is obtained, the study personnel at each participating center will add the patient to a ICF log (spreadsheet) and attribute a study number to each participant. The hospital study personnel will assign a specific patient access card to the participant and register its code on the ICF log. Data entered into the App and transferred to the sponsor's database will thus be fully anonymized.

The ICF log will allow the hospital study personnel to reconcile data with individual patient identity and should be kept by hospital study personnel in a secured location. Therefore, only the medical staff under the responsibility of the investigator in each participating center will be able to establish a link between the identity of the patient and the data collected throughout the study. The ICF log will not be communicated to the sponsor.

For the statistical analysis, the scientific staff of the Heart Centre Hasselt will only receive and process anonymized data. The generation of anonymous patient code is done via a Universally Unique Identifier (UUID), a 128-bit label generated according to standard methods that guarantee the uniqueness and the non-reversibility. Therefore, the Heart Centre Hasselt will not process any personal data and is therefore not subject to GDPR requirements.

Smartphone intervention:

Personalized alarm limits that can be predefined include:

* Heart rate: an upper rate will be set to detect possible atrial fibrillation
* Weight gain: ideal weight and alarm weight can be set by the case nurse.
* Blood pressure: hypotension (under normal limits for the specific patient) and extreme hypertension.
* Not using the application, no measurement input by the patient for a predefined time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HF - NYHA class II-IV
* LVEF ≤50%.
* Hospitalisation due to decompensated HF at the moment of inclusion or up to 1 month prior to inclusion (i.e. discharged ≤1 month prior to inclusion).
* Owning a smartphone and able to use an application
* Written informed consent obtained

Exclusion Criteria:

* Acute coronary syndrome
* High urgent listed for heart transplantation
* Planned revascularisation, TAVI, MitraClip and/or CRT implantation within 3 months after inclusion
* Known alcohol or drug abuse
* Terminal renal insufficiency with haemodialysis or peritoneal dialysis
* Impairment or unwillingness to use the digital support equipment (e.g. dementia, impaired self-determination, lacking ability to communicate)
* Existence of any non-cardiac disease reducing life expectancy to less than 1 year
* Age <18 years
* Participation in other treatment studies or remote patient management programmes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-05-21 (Actual); Primary Completion 2022-11-21 (Estimated); Study Completion 2022-11-21 (Estimated)

PRIMARY OUTCOMES:
Efficiency measures | Through study completion, an average of 6 months
  Demonstrate that this solution makes good use of time and energy in a way that does not waste it.
  This will be measured via daily time spent by case nurses using the platform, compared to time spent without the solution.
Cost-effectiveness | Through study completion, an average of 6 months
  To evaluate the implementation cost of the system, and to demonstrate cost-effectiveness. It will be calculated using healthcare cost data and work productivity and impairment (WPAI) questionnaire to calculate incremental cost-effectiveness ratio (ICER).

SECONDARY OUTCOMES:
Patient acceptability | at 3 and 6 months
  SUTAQ (Service User Technology Acceptability Questionnaire)
Adoption and sustainability | Through study completion, an average of 6 months
  Average created between the number of patients refusing inclusion, patients who dropped out before the end of the study, and patients continuing to use the application during the 6 months.
Quality of patient life | At the recruitment, after 3 ans 6 months
  MLHFQ (Minnesota living with heart failure questionnaire): comparison between the patient's quality of life with and without the tool
Patient literacy | At the recruitment, after 3 ans 6 months
  HLS-EU-Q16 (European Health literacy Questionnaire): comparison between patient literacy at recruitment and at the end of the study
Patient self-care | At the recruitment, after 3 ans 6 months
  EHFScB-9 (The European Heart Failure Self-care Behaviour scale): comparison between the self-care patient at recruitment and at the end of the study
The rate of unplanned cardiovascular readmission/mortality | Through study completion, an average of 6 months
  The difference between the rate of unplanned cardiovascular readmission/mortality in patients with and without the app.

CONTACTS AND LOCATIONS:
Locations (1):
- Attipoe, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Abraham WT, Stevenson LW, Bourge RC, Lindenfeld JA, Bauman JG, Adamson PB; CHAMPION Trial Study Group. Sustained efficacy of pulmonary artery pressure to guide adjustment of chronic heart failure therapy: complete follow-up results from the CHAMPION randomised trial. Lancet. 2016 Jan 30;387(10017):453-61. doi: 10.1016/S0140-6736(15)00723-0. Epub 2015 Nov 9. PMID 26560249
- [Background] Hindricks G, Taborsky M, Glikson M, Heinrich U, Schumacher B, Katz A, Brachmann J, Lewalter T, Goette A, Block M, Kautzner J, Sack S, Husser D, Piorkowski C, Sogaard P; IN-TIME study group*. Implant-based multiparameter telemonitoring of patients with heart failure (IN-TIME): a randomised controlled trial. Lancet. 2014 Aug 16;384(9943):583-590. doi: 10.1016/S0140-6736(14)61176-4. PMID 25131977
- [Background] Stehlik J, Schmalfuss C, Bozkurt B, Nativi-Nicolau J, Wohlfahrt P, Wegerich S, Rose K, Ray R, Schofield R, Deswal A, Sekaric J, Anand S, Richards D, Hanson H, Pipke M, Pham M. Continuous Wearable Monitoring Analytics Predict Heart Failure Hospitalization: The LINK-HF Multicenter Study. Circ Heart Fail. 2020 Mar;13(3):e006513. doi: 10.1161/CIRCHEARTFAILURE.119.006513. Epub 2020 Feb 25. PMID 32093506
- [Background] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Kirwan BA, Winkler S, Vettorazzi E, Bruch L, Oeff M, Zugck C, Doerr G, Naegele H, Stork S, Butter C, Sechtem U, Angermann C, Gola G, Prondzinsky R, Edelmann F, Spethmann S, Schellong SM, Schulze PC, Bauersachs J, Wellge B, Schoebel C, Tajsic M, Dreger H, Anker SD, Stangl K. Efficacy of telemedical interventional management in patients with heart failure (TIM-HF2): a randomised, controlled, parallel-group, unmasked trial. Lancet. 2018 Sep 22;392(10152):1047-1057. doi: 10.1016/S0140-6736(18)31880-4. Epub 2018 Aug 25. PMID 30153985
- [Background] Keutzer L, Simonsson US. Medical Device Apps: An Introduction to Regulatory Affairs for Developers. JMIR Mhealth Uhealth. 2020 Jun 26;8(6):e17567. doi: 10.2196/17567. PMID 32589154
- [Background] Urbich M, Globe G, Pantiri K, Heisen M, Bennison C, Wirtz HS, Di Tanna GL. A Systematic Review of Medical Costs Associated with Heart Failure in the USA (2014-2020). Pharmacoeconomics. 2020 Nov;38(11):1219-1236. doi: 10.1007/s40273-020-00952-0. PMID 32812149
- [Background] Lesyuk W, Kriza C, Kolominsky-Rabas P. Cost-of-illness studies in heart failure: a systematic review 2004-2016. BMC Cardiovasc Disord. 2018 May 2;18(1):74. doi: 10.1186/s12872-018-0815-3. PMID 29716540
- [Background] Ware P, Ross HJ, Cafazzo JA, Laporte A, Seto E. Implementation and Evaluation of a Smartphone-Based Telemonitoring Program for Patients With Heart Failure: Mixed-Methods Study Protocol. JMIR Res Protoc. 2018 May 3;7(5):e121. doi: 10.2196/resprot.9911. PMID 29724704
- [Background] Ware P, Ross HJ, Cafazzo JA, Boodoo C, Munnery M, Seto E. Outcomes of a Heart Failure Telemonitoring Program Implemented as the Standard of Care in an Outpatient Heart Function Clinic: Pretest-Posttest Pragmatic Study. J Med Internet Res. 2020 Feb 8;22(2):e16538. doi: 10.2196/16538. PMID 32027309
- See also: Comunicare - Care companion. Comunicare connects the patient with his/her care givers. (Website of the device under study) — http://www.comunicare.be/

DOCUMENTS (1):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT05487365/Prot_000.pdf